CLINICAL TRIAL: NCT04976855
Title: A Phase I Double-Blind, Placebo-Controlled Randomized Study to Assess Repeated Doses of INDV-2000 (C4X_3256) up to 28 Days in Healthy Volunteers, and an Open-Label Study of INDV-2000 up to 11 Days in Treatment Seeking Individuals With Opioid Use Disorder
Brief Title: Study to Assess Repeated Doses of INDV-2000 in Healthy Volunteers and in Treatment Seeking Individuals With Opioid Use Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: INDV-2000-102; UG3DA050308 (NIH)
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteer; Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part I Cohort 1 INDV-2000 100 mg QD (Experimental): Healthy volunteers will receive INDV-2000 100 mg once daily for 7 days.
  Interventions: Drug: INDV-2000
- Part I Cohort 1 Placebo (Placebo Comparator): Healthy volunteers will receive placebo once daily for 7 days.
  Interventions: Drug: Placebo
- Part I Cohort 2 INDV-2000 100 mg BID (Experimental): Healthy volunteers will receive INDV-2000 100 mg twice daily for 7 days.
  Interventions: Drug: INDV-2000
- Part I Cohort 2 Placebo (Placebo Comparator): Healthy volunteers will receive placebo twice daily for 7 days.
  Interventions: Drug: Placebo
- Part II Cohort 1 INDV-2000 200 mg BID (Experimental): Healthy volunteers will receive INDV-2000 200 mg twice daily for 28 days.
  Interventions: Drug: INDV-2000
- Part II Cohort 1 Placebo (Placebo Comparator): Healthy volunteers will receive placebo twice daily for 28 days.
  Interventions: Drug: Placebo
- Part II Cohort 2 INDV-2000 400 mg BID (Experimental): Healthy volunteers will receive INDV-2000 400 mg twice daily for 28 days.
  Interventions: Drug: INDV-2000
- Part II Cohort 2 Placebo (Placebo Comparator): Healthy volunteers will receive placebo twice daily for 28 days.
  Interventions: Drug: Placebo
- Part III INDV-2000 400 mg BID + SUBOXONE SL Film (Experimental): Participants with opioid use disorder will receive SUBOXONE sublingual (SL) film for 6 days during the run-in period. Participants will then receive SUBOXONE SL film alone for 2 days, then SUBOXONE SL film and INDV-2000 for 7 days followed by INDV-2000 dosing alone for 4 days.
  Interventions: Drug: INDV-2000; Drug: SUBOXONE® sublingual film

INTERVENTIONS:
Drug: INDV-2000 — Capsule for oral administration
  Other Names: C4X_3256
  Arms: Part I Cohort 1 INDV-2000 100 mg QD; Part I Cohort 2 INDV-2000 100 mg BID; Part II Cohort 1 INDV-2000 200 mg BID; Part II Cohort 2 INDV-2000 400 mg BID; Part III INDV-2000 400 mg BID + SUBOXONE SL Film
Drug: Placebo — Capsule for oral administration
  Arms: Part I Cohort 1 Placebo; Part I Cohort 2 Placebo; Part II Cohort 1 Placebo; Part II Cohort 2 Placebo
Drug: SUBOXONE® sublingual film — Administered either under the tongue (sublingual) or between the gum and cheek (buccal)
  Other Names: Buprenorphine and naloxone
  Arms: Part III INDV-2000 400 mg BID + SUBOXONE SL Film

SUMMARY:
The primary objectives for the study are:

* Part I and Part II: Assess safety and tolerability of repeated doses of INDV-2000 in healthy volunteers.
* Part III: Assess the safety and tolerability of repeated doses of INDV-2000 administered alone and with SUBOXONE sublingual (SL) film in an opioid use disorder (OUD) treatment seeking population.

DETAILED DESCRIPTION:
The study will be conducted in 3 parts:

Part I: Double-blind, placebo-controlled, randomized, multiple ascending dose study for 7 days of dosing with INDV-2000 in healthy volunteers.

Part II: Double-blind, placebo-controlled, randomized, multiple ascending dose study for 28 days of dosing with INDV-2000 in healthy volunteers.

Part III: This part is an open-label study in OUD treatment seeking individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Able to verbalize understanding of the consent form, able to provide written informed consent, and verbalize willingness to complete study procedures, be able to comply with protocol requirements, rules and regulations of study site, and be likely to complete all the study interventions.
2. Female subjects of child-bearing potential who are sexually active with males must use, with their partner, a condom plus an approved method of effective contraception from the time of screening until 30 days after the last dose of Investigational Medicinal Product (IMP). The impact of IMP on the efficacy of hormonal contraceptives is unknown. Male subjects who are sexually active with female partners of child-bearing potential must use, with their partner, a condom plus an approved method of effective contraception from the time of screening until 90 days after the last dose of IMP and agree to not donate sperm over this time period. Effective methods of contraception are:

   1. Combined (estrogen and progestogen-containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, or transdermal
   2. Progestogen-only hormonal contraception: oral, injectable/implantable, or intrauterine hormone-releasing system (IUD)
   3. Implantable intrauterine device (IUS)
   4. Surgical sterilization (for example, vasectomy or bilateral tubal ligation)
   5. Male condom with spermicidal gel/foam or with female cap or diaphragm (double barrier)
   6. abstinence from heterosexual intercourse as a conscious choice and established pattern of lifestyle

   Part I and II only:
3. Healthy male or female.
4. Between 18 and 55 years of age inclusive.
5. Body mass index (BMI) within 18.0 to 32.0 kg/m^2, inclusive (minimum weight of at least 50.0 kg at Screening).

   Part III only:
6. Male or female seeking treatment for OUD with a diagnosis of moderate or severe OUD by Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria.
7. Between 18 and 65 years of age inclusive.
8. BMI within 18.0 to 35.0 kg/m^2, inclusive (minimum weight of at least 50.0 kg at Screening).

Exclusion Criteria:

1. Have a medical history of clinically significant neurological, cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, or psychiatric disorder as judged by an Investigator.
2. Have clinically significant abnormal biochemistry, hematology or urinalysis results as judged by an Investigator or medically responsible physician.
3. Have a history of narcolepsy or other significant sleep disorders.
4. Have disorders that may interfere with drug absorption, distribution, metabolism and excretion (ADME) processes.
5. Positive test results for human immunodeficiency virus (HIV)-1/HIV-2 antibodies, hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCVAb).
6. Serious cardiac illness or other cardiac assessments including, but not limited to:

   1. Uncontrolled arrhythmias.
   2. History of congestive heart failure (CHF).
   3. Myocardial infarction <6 months from receipt of first dose of IMP
   4. Uncontrolled symptomatic angina
   5. QTcF > 450 msec for males and > 470 msec for females or history of prolonged QT syndrome.
7. Current active hepatic or biliary disease, including subjects with cholecystectomy <90 days prior to Screening.
8. Concurrent treatment or treatment with an investigational drug within 30 days prior to the first dose of any study drug.
9. History of suicidal ideation within 30 days prior to providing written informed consent as evidenced by answering "yes' to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) completed at the Screening Visit or history of a suicide attempt (per the C-SSRS) in the 6 months prior to informed consent.
10. Pregnant or lactating females.
11. Any consumption of food or drink containing poppy seeds, grapefruit or Seville oranges within 7 days prior to the IMP administration.
12. Treatment with any known drugs that are moderate or strong inhibitors/inducers of cytochrome P450 (CYP) 3A4 within 30 days prior to first dose of IMP.
13. Known allergy or hypersensitivity to IMP or its excipients.
14. Any condition that, in the opinion of an Investigator or medically responsible physician, would interfere with evaluation of the IMP or interpretation of subject safety or study results.
15. Affiliated with, or a family member of, site staff directly involved in the study, or anyone with a financial interest in the outcome of the study.
16. Subjects who are unable, in the opinion of an Investigator or medically responsible physician, to comply fully with the study requirements.
17. Participation in any other clinical study within 30 days prior to signing the informed consent form.
18. Current incarceration or pending incarceration/legal action that could prevent participation or compliance in the study.

    Part I and II only:
19. Regular alcohol consumption in males > 21 units per week and females > 14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine).
20. Positive test result for alcohol and/or any drugs of abuse at screening
21. Have a blood pressure reading outside of the following range: Systolic < 86 or > 149 mmHg; Diastolic < 50 or > 94 mmHg
22. Current smokers and those who have smoked within the last 90 days. Current users of e-cigarettes and nicotine replacement products, and those who have used these products within the last 90 days.
23. Blood donation of greater than 500 mL within 56 days or plasma donation within 7 days of screening; clinically significant anemia or low hemoglobin (<11 g/dL for females, <12 g/dL for males).
24. Healthy volunteers who are taking, or have taken, any prescribed or over-the-counter drugs (other than 2 g per day acetaminophen, hormone replacement therapy [HRT], hormonal contraception) or herbal remedies in the 14 days before IMP administration. Exceptions may apply on a case by case basis if considered not to interfere with the objectives of the study, as agreed by an Investigator and Sponsor's Medical Monitor.

    Part III only:
25. Regular alcohol consumption in males > 27 units per week and females > 20 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine).
26. Current substance use disorder, as defined by DSM-5 criteria, with any substances other than opioids, tobacco, cannabis, or alcohol, or dependence with any substance that would interfere with the completion of the study by judgment of the Investigator or medically responsible physician.
27. Current history of alcohol withdrawal within one year prior to screening.
28. Blood donation of greater than 500 mL within 56 days or plasma donation within 7 days of screening; clinically significant anemia or low hemoglobin (< 10 g/dL for females, < 12 g/dL for males).
29. Have a blood pressure reading outside of the following range: Systolic < 86 or > 159 mmHg; Diastolic < 50 or > 99 mmHg. Investigator should rule out acute changes resulting from opioid withdrawal.
30. Has total bilirubin ≥ 1.5 × upper limit of normal (ULN) (with direct bilirubin > 1.3 mg/dL), alanine aminotransferase (ALT) ≥ 3 × ULN, aspartate aminotransferase (AST) ≥ 3 × ULN, serum creatinine > 2 × ULN, or international normalized ratio (INR) > 1.5 × ULN at Screening).
31. Received medication-assisted treatment for OUD (e.g., methadone, buprenorphine) in the 30 days prior to providing written informed consent.
32. Received any prior treatment with a buprenorphine implant or injection.
33. Treatment for OUD required by court order.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Johns Hopkins University School of Medicine BPRU, Baltimore, Maryland
  - InSite Clinical Research, DeSoto, Texas
  - Worldwide Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in 3 parts: Part I and Part II in healthy volunteers, and Part III in treatment seeking individuals with opioid use disorder (OUD).
Groups:
- Part I: INDV-2000 100 mg QD: Healthy volunteers received INDV-2000 once daily for 7 days.
  INDV-2000: 100 mg/capsule for oral administration
- Part I: INDV-2000 100 mg BID: Healthy volunteers received INDV-2000 twice daily for 7 days.
  INDV-2000: 100 mg/capsule for oral administration
- Part I: Placebo (Pooled): Healthy volunteers received placebo either once daily or twice daily for 7 days.
  Placebo: Capsule for oral administration
- Part II: INDV-2000 200 mg BID: Healthy volunteers received INDV-2000 twice daily for 28 days.
  INDV-2000: One 200 mg/capsule for oral administration
- Part II: INDV-2000 400 mg BID: Healthy volunteers received INDV-2000 twice daily for 28 days.
  INDV-2000: Two 200 mg/capsule for oral administration
- Part II: Placebo (Pooled): Healthy volunteers received placebo twice daily for 28 days.
  Placebo: Either one or two capsules for oral administration
- Part III: INDV-2000 400 mg BID + SUBOXONE SL: A single cohort of treatment seeking participants with opioid use disorder (OUD) received SUBOXONE sublingual (SL) film for 6 days during the run-in period. Participants then received SUBOXONE SL film alone on Days 1 and 2, then SUBOXONE SL film and INDV-2000 on Days 3-9, followed by INDV-2000 alone on Days 10-13.
  INDV-2000: Two 200 mg/capsule for oral administration
  SUBOXONE® sublingual film: Administered either under the tongue (sublingual) or between the gum and cheek (buccal)
Period: Part I
Arm/Group | Part I: INDV-2000 100 mg QD | Part I: INDV-2000 100 mg BID | Part I: Placebo (Pooled) | Part II: INDV-2000 200 mg BID | Part II: INDV-2000 400 mg BID | Part II: Placebo (Pooled) | Part III: INDV-2000 400 mg BID + SUBOXONE SL
Started | 9 | 9 | 6 | 0 (Only Part I is reported in this section) | 0 (Only Part I is reported in this section) | 0 (Only Part I is reported in this section) | 0 (Only Part I is reported in this section)
Completed | 9 | 8 | 6 | 0 (Only Part I is reported in this section) | 0 (Only Part I is reported in this section) | 0 (Only Part I is reported in this section) | 0 (Only Part I is reported in this section)
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part II
Arm/Group | Part I: INDV-2000 100 mg QD | Part I: INDV-2000 100 mg BID | Part I: Placebo (Pooled) | Part II: INDV-2000 200 mg BID | Part II: INDV-2000 400 mg BID | Part II: Placebo (Pooled) | Part III: INDV-2000 400 mg BID + SUBOXONE SL
Started | 0 (Only Part II is reported in this section) | 0 (Only Part II is reported in this section) | 0 (Only Part II is reported in this section) | 9 | 9 | 6 | 0 (Only Part II is reported in this section)
Completed | 0 (Only Part II is reported in this section) | 0 (Only Part II is reported in this section) | 0 (Only Part II is reported in this section) | 8 | 8 | 5 | 0 (Only Part II is reported in this section)
Not Completed | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Part III: Run-in Period (6 Days)
Arm/Group | Part I: INDV-2000 100 mg QD | Part I: INDV-2000 100 mg BID | Part I: Placebo (Pooled) | Part II: INDV-2000 200 mg BID | Part II: INDV-2000 400 mg BID | Part II: Placebo (Pooled) | Part III: INDV-2000 400 mg BID + SUBOXONE SL
Started | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 16
Completed | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part III: Treatment Period (14 Days)
Arm/Group | Part I: INDV-2000 100 mg QD | Part I: INDV-2000 100 mg BID | Part I: Placebo (Pooled) | Part II: INDV-2000 200 mg BID | Part II: INDV-2000 400 mg BID | Part II: Placebo (Pooled) | Part III: INDV-2000 400 mg BID + SUBOXONE SL
Started | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 16
Completed | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 0 (Only Part III is reported in this section) | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population for Part I, Part II and Part III, defined as participants who received at least 1 dose of INDV-2000.
Groups:
- Part III: INDV-2000 400 mg BID + SUBOXONE SL: A single cohort of treatment seeking participants with opioid use disorder (OUD) received SUBOXONE sublingual (SL) film for 6 days during the run-in period. Participants then received SUBOXONE SL film alone for 2 days, then SUBOXONE SL film and INDV-2000 for 7 days, followed by INDV-2000 dosing alone for 4 days.
  INDV-2000: Two 200 mg/capsule for oral administration
  SUBOXONE® sublingual film: Administered either under the tongue (sublingual) or between the gum and cheek (buccal)
- Total: Total of all reporting groups
Arm/Group | Part I: INDV-2000 100 mg QD | Part I: INDV-2000 100 mg BID | Part I: Placebo (Pooled) | Part II: INDV-2000 200 mg BID | Part II: INDV-2000 400 mg BID | Part II: Placebo (Pooled) | Part III: INDV-2000 400 mg BID + SUBOXONE SL | Total
Number analyzed (Participants) | 9 | 9 | 6 | 9 | 9 | 6 | 16 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (11.29) | 38.3 (6.50) | 36.7 (11.48) | 40.2 (8.17) | 40.6 (9.00) | 35.7 (11.31) | 39.9 (4.89) | 39.1 (8.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 1 | 3 | 0 | 4 | 12
  Male | 7 | 8 | 5 | 8 | 6 | 6 | 12 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 3 | 7 | 5 | 2 | 5 | 32
  White | 4 | 4 | 2 | 1 | 4 | 4 | 11 | 30
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 6 | 9 | 9 | 6 | 16 | 64
Weight [Mean (Standard Deviation); unit: kg] | 78.18 (10.103) | 82.67 (11.630) | 86.20 (15.129) | 76.48 (5.833) | 82.00 (16.252) | 82.25 (13.536) | 86.24 (19.333) | 82.26 (14.226)

OUTCOME MEASURES:

1. Primary Outcome: Part I and Part II: Number of Participants With Adverse Events
Time Frame: From first dose of study drug up to 7 days after last dose (up to 14 days in Part I and 35 days in Part II).
Measure: Number; unit: Participants
Arm/Group | Part I: INDV-2000 100 mg QD | Part I: INDV-2000 100 mg BID | Part I: Placebo (Pooled) | Part II: INDV-2000 200 mg BID | Part II: INDV-2000 400 mg BID | Part II: Placebo (Pooled)
Number analyzed (Participants) | 9 | 9 | 6 | 9 | 9 | 6
Participants
  Any TEAE | 5 | 2 | 3 | 8 | 8 | 2
  Serious | 1 | 0 | 0 | 0 | 0 | 0
  Study drug-related | 5 | 0 | 2 | 8 | 6 | 1
  Serious and Study drug-related | 0 | 0 | 0 | 0 | 0 | 0
  Severe | 1 | 0 | 0 | 0 | 0 | 0
  Discontinuation | 0 | 0 | 0 | 1 | 0 | 1
  Death | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part III: Number of Participants With Adverse Events
Time Frame: From first dose of INDV-2000 up to 7 days after last dose (up to 18 days).
Measure: Count of Participants; unit: Participants
Arm/Group | Part III: INDV-2000 400 mg BID + SUBOXONE SL
Number analyzed (Participants) | 16
Participants
  Any TEAE | 5
  Serious | 0
  Study-drug related | 2
  Serious and Study-drug related | 0
  Severe | 0
  Discontinuation | 0
  Death | 0

3. Secondary Outcome: Part I and Part II: Maximum Plasma Concentration (Cmax) of INDV-2000 Following Dosing on Days 1 and 7 for Part I and Days 1, 7, and 28 for Part II
Description: Day 28 is only for Part II.
Time Frame: Days 1 and 7 for Part I and Days 1, 7, and 28 for Part II, predose and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part I: INDV-2000 100 mg QD | Part I: INDV-2000 100 mg BID | Part II: INDV-2000 200 mg BID | Part II: INDV-2000 400 mg BID
Number analyzed (Participants) | 9 | 9 | 9 | 9
ng/mL
  Day 1 | 849 (51.9) | 759 (36.3) | 1480 (50.1) | 1830 (43.8)
  Day 7 | 967 (34.3) | 855 (32.6) | 1570 (49.0) | 1670 (45.2)
  Day 28: number analyzed (Participants) | 0 | 0 | 9 | 9
  Day 28 |  |  | 1780 (40.0) | 1920 (36.2)

4. Secondary Outcome: Part I and Part II: Time to Maximum Plasma Concentration (Tmax) of INDV-2000 Following Dosing on Days 1 and 7 for Part I and Days 1, 7, and 28 for Part II
Description: Day 28 is only for Part II
Time Frame: as for outcome 3
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: hour
Arm/Group | Part I: INDV-2000 100 mg QD | Part I: INDV-2000 100 mg BID | Part II: INDV-2000 200 mg BID | Part II: INDV-2000 400 mg BID
Number analyzed (Participants) | 9 | 9 | 9 | 9
hour
  Day 1 | 4 [2 to 8] | 2 [2 to 8] | 3 [2 to 6] | 2 [2 to 4]
  Day 7 | 3 [2 to 6] | 1 [1 to 4] | 4 [2 to 6] | 2 [1 to 4]
  Day 28: number analyzed (Participants) | 0 | 0 | 9 | 9
  Day 28 |  |  | 2 [1 to 4] | 2 [2 to 4]

5. Secondary Outcome: Part I and Part II: Area Under the Plasma Concentration-time Curve (AUC0-τ) of INDV-2000 Following Dosing on Days 1 and 7 for Part I and Days 1, 7, and 28 for Part II
Description: τ = 12 hours for BID dosing and 24 hours for QD dosing. Day 28 is only for Part II.
Time Frame: as for outcome 3
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Part I: INDV-2000 100 mg QD | Part I: INDV-2000 100 mg BID | Part II: INDV-2000 200 mg BID | Part II: INDV-2000 400 mg BID
Number analyzed (Participants) | 9 | 9 | 9 | 9
hour*ng/mL
  Day 1, AUC0-τ | 5800 (64.4) | 4760 (31.8) | 9460 (34.7) | 11900 (44.9)
  Day 7, AUC0-τ | 5660 (56.8) | 5570 (26.7) | 8930 (43.2) | 12000 (43.2)
  Day 28, AUC0-τ: number analyzed (Participants) | 0 | 0 | 9 | 9
  Day 28, AUC0-τ |  |  | 11600 (42.0) | 12700 (31.4)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 7 days after last dose (up to 14 days in Part I and 35 days in Part II). From first dose of INDV-2000 up to 7 days after last dose (up to 18 days) in Part III.
Arm/Group | Part I: INDV-2000 100 mg QD | Part I: INDV-2000 100 mg BID | Part I: Placebo (Pooled) | Part II: INDV-2000 200 mg BID | Part II: INDV-2000 400 mg BID | Part II: Placebo (Pooled) | Part III: INDV-2000 400 mg BID + SUBOXONE SL
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/6 | 0/9 | 0/9 | 0/6 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/9 | 0/6 | 0/9 | 0/9 | 0/6 | 0/16
Other Adverse Events (participants affected / at risk) | 5/9 | 2/9 | 3/6 | 8/9 | 8/9 | 2/6 | 5/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part I: INDV-2000 100 mg QD (N=9) | Part I: INDV-2000 100 mg BID (N=9) | Part I: Placebo (Pooled) (N=6) | Part II: INDV-2000 200 mg BID (N=9) | Part II: INDV-2000 400 mg BID (N=9) | Part II: Placebo (Pooled) (N=6) | Part III: INDV-2000 400 mg BID + SUBOXONE SL (N=16)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: INDV-2000 100 mg QD (N=9) | Part I: INDV-2000 100 mg BID (N=9) | Part I: Placebo (Pooled) (N=6) | Part II: INDV-2000 200 mg BID (N=9) | Part II: INDV-2000 400 mg BID (N=9) | Part II: Placebo (Pooled) (N=6) | Part III: INDV-2000 400 mg BID + SUBOXONE SL (N=16)
Somnolence (Nervous system disorders) | 5 | 0 | 2 | 8 | 6 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 2 | 1 | 1 | 0
Dizzines (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0
Vessel puncture site pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dental paraesthesia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lacerations (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feces discolored (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT04976855/Prot_000.pdf
  • Statistical Analysis Plan: Parts I & II (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT04976855/SAP_001.pdf
  • Statistical Analysis Plan: Part III (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT04976855/SAP_002.pdf